CLINICAL TRIAL: NCT00004054
Title: A Phase III Protocol of Androgen Suppression (AS) and Radiation Therapy (RT) vs AS and RT Followed by Chemotherapy With Paclitaxel, Estramustine, and Etoposide (TEE) for Localized, High-Risk, Prostate Cancer
Brief Title: Hormone Therapy Plus Radiation Therapy With or Without Combination Chemotherapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9902; CDR0000067250
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Estramustine; Etoposide; Flutamide; Paclitaxel; Gonadotropin-Releasing Hormone; Radiotherapy; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hormones and RT (Experimental): Androgen suppression (AS) (Luteinizing hormone releasing hormone agonist and bicalutamide [Casodex] or flutamide [Eulexin]) x 8 weeks followed by RT to 70.2 Gy with concurrent AS (LHRH agonist and bicalutamide [Casodex] or flutamide [Eulexin]). AS will continue for a total of 24 months from initiation of all treatment. Oral anti-androgen will be discontinued at the end of radiation therapy (RT).
  Interventions: Drug: bicalutamide; Drug: flutamide; Drug: Luteinizing hormone releasing hormone [LHRH] agonist; Radiation: Radiation therapy
- Hormones and RT plus Chemotherapy (Experimental): AS (LHRH agonist and bicalutamide [Casodex] or flutamide [Eulexin]) x 8 weeks followed by RT to 70.2 Gy with concurrent AS (LHRH agonist and bicalutamide [Casodex] or flutamide [Eulexin]) and estramustine phosphate sodium, etoposide, paclitaxel, and warfarin [Coumadin®]. AS will continue for a total of 24 months from initiation all treatment. Oral antiandrogen will be discontinued at the end of RT.
  Interventions: Drug: bicalutamide; Drug: estramustine phosphate sodium; Drug: etoposide; Drug: flutamide; Drug: paclitaxel; Radiation: Radiation therapy; Drug: warfarin

INTERVENTIONS:
Drug: bicalutamide — Administered orally at a dose of one 50mg tablet per day. Begins 8 weeks prior to radiotherapy and continues throughout radiotherapy.
  Other Names: Casodex
Drug: estramustine phosphate sodium — 280 mg three times a day for 14 days and repeated every 3 weeks for 4 cycles
  Arms: Hormones and RT plus Chemotherapy
Drug: etoposide — 50 mg/m^2 in divided doses b.i.d. for 14 days and repeated every 3 weeks for 4 cycles
  Arms: Hormones and RT plus Chemotherapy
Drug: flutamide — Administered orally at a dose of two 125 mg capsules three times a day for a total daily dose of 750 mg. Begins 8 weeks prior to radiotherapy and continues throughout radiotherapy.
  Other Names: Eulexin
Drug: paclitaxel — 135 mg/m^2 given as a 1-hour infusion (on day 2 of each cycle) and repeated every 3 weeks for 4 cycles
  Arms: Hormones and RT plus Chemotherapy
Drug: Luteinizing hormone releasing hormone [LHRH] agonist — Releasing hormone agonists (such as leuprolide, goserelin, buserelin, triptorelin) will be given for 4 months
  Arms: Hormones and RT
Radiation: Radiation therapy — Radiation will begin 8 weeks following the initiation of hormone administration: 46.8 Gy to the regional lymphatics followed by a 23.4 Gy boost to the prostate to bring the total dose to the prostate to 70.2 Gy. Daily tumor doses will be 1.8 Gy per day, 5 days per week x 7-8 weeks.
Drug: warfarin — To keep international normalized ratio (INR) > 1.5 and < 2.5; begins with the start of chemotherapy and will be given continuously until 4 weeks after the end of the fourth cycle of chemotherapy
  Other Names: Coumadin
  Arms: Hormones and RT plus Chemotherapy

SUMMARY:
RATIONALE: Hormones can stimulate the production of prostate cancer cells. Hormone therapy may fight prostate cancer by reducing the production of androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether hormone therapy plus radiation therapy is more effective with or without combination chemotherapy for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of hormone therapy plus radiation therapy with or without combination chemotherapy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of androgen suppression and radiotherapy with or without subsequent paclitaxel, estramustine, and etoposide, in terms of overall and disease-free survival, biochemical and local control, and freedom from distant metastasis, in patients with localized high-risk prostate cancer.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to prostate-specific antigen level (≤ 10 ng/mL vs 11-100 ng/mL), tumor stage (T1-2 vs T3-4), Gleason score (7 vs 8-10), and prior hormone use (yes vs no). Patients are randomized to one of two treatment arms.

All patients receive androgen suppression comprising a luteinizing hormone-releasing hormone (LHRH) agonist AND bicalutamide OR flutamide for 4 months. Beginning 8 weeks after the initiation of androgen suppression, all patients undergo radiotherapy once daily, 5 days a week, for 7-8 weeks. Patients who received prior androgen suppression therapy count time to radiotherapy from start date of prior hormonal therapy.

* Arm I: Patients continue androgen suppression therapy (LHRH agonist only) for approximately 20 more months after radiotherapy is completed.
* Arm II: Patients continue therapy as in arm I and receive chemotherapy beginning 28 days after completing radiotherapy. Chemotherapy comprises oral estramustine 3 times daily and oral etoposide twice daily on days 1-14 and paclitaxel IV over 1 hour on day 2. Chemotherapy repeats every 21 days for 4 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,440 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven prostate cancer at high risk for relapse as determined by either of the following:

  * Prostate-specific antigen (PSA) 20-100 ng/mL and Gleason score at least 7 (any T stage)
  * Clinical stage at least T2, Gleason score at least 8, and PSA no greater than 100 ng/mL
* Negative lymph nodes
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Zubrod 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* White blood cell (WBC) count of at least 3,000/mm^3
* Platelet count at least 130,000/mm^3
* Hemoglobin at least 11.4 g/dL

Hepatic:

* Aspartate aminotransferase (AST) no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.5 mg/dL

Other:

* No other invasive cancer within the past 5 years except superficial nonmelanomatous skin cancer
* No major medical or psychiatric illness that would preclude study participation
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 5 years since prior chemotherapy

Endocrine therapy:

* At least 60 days since prior finasteride for prostatic hypertrophy
* At least 90 days since prior testosterone
* No more than 30 days since initiation of prior pharmacologic androgen ablation for prostate cancer

Radiotherapy:

* No prior pelvic radiotherapy
* No concurrent intensity-modulated radiotherapy

Surgery:

* No prior radical prostatectomy
* No prior cryosurgery for prostate cancer
* No prior orchiectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2000-01; Primary Completion 2010-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M. Sandler, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (54):
- United States (52):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Baptist Hospital of Miami, Miami, Florida
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
- Canada (2):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario

REFERENCES:
- [Result] Rosenthal SA, Bae K, Pienta KJ, Sobczak ML, Asbell SO, Rajan R, Kerlin KJ, Michalski JM, Sandler HM; Radiation Therapy Oncology Group Trial 9902. Phase III multi-institutional trial of adjuvant chemotherapy with paclitaxel, estramustine, and oral etoposide combined with long-term androgen suppression therapy and radiotherapy versus long-term androgen suppression plus radiotherapy alone for high-risk prostate cancer: preliminary toxicity analysis of RTOG 99-02. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):672-8. doi: 10.1016/j.ijrobp.2008.05.020. Epub 2008 Nov 5. PMID 18990504
- [Result] Rosenthal SA, Hunt D, Sartor AO, Pienta KJ, Gomella L, Grignon D, Rajan R, Kerlin KJ, Jones CU, Dobelbower M, Shipley WU, Zeitzer K, Hamstra DA, Donavanik V, Rotman M, Hartford AC, Michalski J, Seider M, Kim H, Kuban DA, Moughan J, Sandler H. A Phase 3 Trial of 2 Years of Androgen Suppression and Radiation Therapy With or Without Adjuvant Chemotherapy for High-Risk Prostate Cancer: Final Results of Radiation Therapy Oncology Group Phase 3 Randomized Trial NRG Oncology RTOG 9902. Int J Radiat Oncol Biol Phys. 2015 Oct 1;93(2):294-302. doi: 10.1016/j.ijrobp.2015.05.024. Epub 2015 Jul 21. PMID 26209502
- [Derived] Nguyen PL, Huang HR, Spratt DE, Davicioni E, Sandler HM, Shipley WU, Efstathiou JA, Simko JP, Pollack A, Dicker AP, Roach M, Rosenthal SA, Zeitzer KL, Mendez LC, Hartford AC, Hall WA, Desai AB, Rabinovitch RA, Peters CA, Rodgers JP, Tran P, Feng FY. Analysis of a Biopsy-Based Genomic Classifier in High-Risk Prostate Cancer: Meta-Analysis of the NRG Oncology/Radiation Therapy Oncology Group 9202, 9413, and 9902 Phase 3 Randomized Trials. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):521-529. doi: 10.1016/j.ijrobp.2022.12.035. Epub 2022 Dec 31. PMID 36596347
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Hormones and RT: Androgen suppression (AS) (Luteinizing hormone releasing hormone [LHRH] agonist and bicalutamide [Casodex] or flutamide [Eulexin]) x 8 weeks followed by RT to 70.2 Gy with concurrent AS (LHRH agonist and bicalutamide [Casodex] or flutamide [Eulexin]). AS will continue for a total of 24 months from initiation of all treatment. Oral anti-androgen will be discontinued at the end of radiation therapy (RT).
Period: Overall Study
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Started | 197 | 200
Completed | 197 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy | Total
Number analyzed (Participants) | 197 | 200 | 397
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 79] | 67 [42 to 81] | 66 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 197 | 200 | 397

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (5-year Rate Reported)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at date of last contact. This analysis was planned to occur when all patients had been potentially followed for 5 years.
Time Frame: From the date of randomization to the date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years.
Population: All randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Number analyzed (Participants) | 197 | 200
percentage of participants | 84.9 [79.9 to 90] | 87.2 [82.4 to 91.9]
Statistical Analysis 1: Comparison: Hormones and RT vs Hormones and RT Plus Chemotherapy; The original target sample size was 1440 patients with a requirement of 340 deaths to test the hypothesis of overall survival (OS) efficacy of the hormones and RT plus chemotherapy arm; the design is based on detecting a 6% absolute improvement in 5-year OS from 79% to 85%, or a 33% relative reduction in the yearly hazard rate, with 90% power and a 2-sided significance level of 0.05; Test type: Superiority or Other; p = 0.81, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.76 to 1.43]

2. Secondary Outcome: Rate of Biochemical Failure at 5 Years
Description: Biochemical failure uses the American Society for Radiation Oncology (ASTRO) definition of prostate-specific antigen (PSA) rises on three consecutive occasions, with biochemical failure date being midway between the last non-rising PSA and the first rise in PSA. Time to biochemical failure is defined as time from randomization to biochemical failure, last known follow-up (censored), or death (competing risk). Biochemical failure rates are estimated using the cumulative incidence method.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been potentially followed for 5 years. Maximum follow-up at time of analysis was 13.3 years.
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Number analyzed (Participants) | 197 | 200
percentage of participants | 48.0 [40.7 to 54.8] | 47.9 [40.7 to 54.8]
Statistical Analysis 1: Comparison: Hormones and RT vs Hormones and RT Plus Chemotherapy; Test type: Superiority; p = 0.82, Gray's test; 2-sided significance level of 0.05; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.74 to 1.27] — Fine-Gray regression model was used to obtain the hazard ratio. Reference level = Hormones and RT

3. Secondary Outcome: Rate of Local Progression at 5 Years
Description: Local progression is defined as documented clinical local and/or regional progression. Time to local progression is defined as time from randomization to local progression, last known follow-up (censored), or death (competing risk). Local progression rates are estimated using the cumulative incidence method.
Time Frame: as for outcome 2
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Number analyzed (Participants) | 197 | 200
percentage of participants | 5.8 [3.1 to 9.7] | 4.1 [1.9 to 7.6]
Statistical Analysis 1: Comparison: Hormones and RT vs Hormones and RT Plus Chemotherapy; Test type: Superiority; p = 0.09, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.28 to 1.10] — Fine-Gray regression model was used to obtain the hazard ratio. Reference level = Hormones and RT

4. Secondary Outcome: Rate of Distant Metastasis at Five Years
Description: Distant metastasis (DM) is defined as documented metastatic disease. Time to distant metastasis is defined as time from randomization to distant metastatic disease, last known follow-up (censored), or death (competing risk). Distant metastasis rates are estimated using the cumulative incidence method.
Time Frame: as for outcome 2
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Number analyzed (Participants) | 197 | 200
percentage of participants | 10.4 [6.6 to 15.2] | 8.3 [4.9 to 12.7]
Statistical Analysis 1: Comparison: Hormones and RT vs Hormones and RT Plus Chemotherapy; Test type: Superiority; p = 0.42, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.48 to 1.36] — Fine-Gray regression model was used to obtain the hazard ratio. Reference level = Hormones and RT

5. Secondary Outcome: Disease-free Survival Rate at 5 Years
Description: Disease-free survival (DFS) was measured from the date of randomization to the date of documentation of progression (local, distant, biochemical failure), death, or last follow-up (censored). The Kaplan-Meier method was used to estimate DFS rates.
Time Frame: as for outcome 2
Population: All randomized patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Number analyzed (Participants) | 197 | 200
percentage of participants | 39.1 [32.2 to 46.0] | 42.9 [35.9 to 49.9]
Statistical Analysis 1: Comparison: Hormones and RT vs Hormones and RT Plus Chemotherapy; Test type: Superiority; p = 0.61, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.19] — Cox proportional hazards model was used to obtain the hazard ratio. Reference level = Hormones and RT

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE).
Groups:
- Hormones and RT: AS (LHRH agonist and Casodex or Eulexin) x 8 weeks followed by RT to 70.2 Gy with concurrent AS (LHRH agonist and Casodex or Eulexin). Androgen suppression will continue for a total of 24 months from initiation of all treatment. Oral anti-androgen will be discontinued at the end of RT.
- Hormones and RT Plus Chemotherapy: AS (LHRH agonist and Casodex or Eulexin) x 8 weeks followed by RT to 70.2 Gy with concurrent AS (LHRH agonist and Casodex or Eulexin) and chemotherapy. Androgen suppression will continue for a total of 24 months from initiation all treatment. Oral antiandrogen will be discontinued at the end of RT.
Arm/Group | Hormones and RT | Hormones and RT Plus Chemotherapy
Serious Adverse Events (participants affected / at risk) | 6/197 | 70/200
Other Adverse Events (participants affected / at risk) | 189/197 | 198/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hormones and RT (N=197) | Hormones and RT Plus Chemotherapy (N=200)
Ferbrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 1
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 0 | 2
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 2 | 11
Esophagitis NOS (Gastrointestinal disorders) | 0 | 1
Late RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 5
Proctitis NOS (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 4
Chest pain (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Pain-other (General disorders) | 0 | 5
Infection NOS (Infections and infestations) | 0 | 2
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 | 2
Infection, Other (Infections and infestations) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Leukopenia NOS (Investigations) | 0 | 23
Neutropenia (Investigations) | 0 | 27
Platelet count decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Secondary malignancy, Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Hematuria present (Renal and urinary disorders) | 0 | 3
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Thrombosis NOS (Vascular disorders) | 0 | 19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hormones and RT (N=197) | Hormones and RT Plus Chemotherapy (N=200)
Hematologic-Other (Blood and lymphatic system disorders) | 1 | 10
Hemoglobin decreased (Blood and lymphatic system disorders) | 23 | 145
Edema NOS (Cardiac disorders) | 7 | 31
Constipation (Gastrointestinal disorders) | 11 | 13
Diarrhea NOS (Gastrointestinal disorders) | 76 | 91
Late RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 54 | 60
Late RT Toxicity: Other GI: NOS (Gastrointestinal disorders) | 23 | 18
Nausea (Gastrointestinal disorders) | 4 | 54
Proctitis NOS (Gastrointestinal disorders) | 42 | 46
Rectal bleeding (Gastrointestinal disorders) | 11 | 9
Stomatitis (Gastrointestinal disorders) | 1 | 10
Vomiting NOS (Gastrointestinal disorders) | 0 | 25
Fatigue (General disorders) | 51 | 110
Late RT Toxicity: Other: NOS (General disorders) | 23 | 18
Pain-other (General disorders) | 14 | 25
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 28 | 23
Alanine aminotransferase increased (Investigations) | 24 | 30
Aspartate aminotransferase increased (Investigations) | 13 | 22
Blood creatinine increased (Investigations) | 5 | 10
Leukopenia NOS (Investigations) | 12 | 98
Lymphopenia (Investigations) | 4 | 15
Neutropenia (Investigations) | 1 | 50
Platelet count decreased (Investigations) | 1 | 31
Prothrombin time prolonged (Investigations) | 0 | 10
Weight decreased (Investigations) | 2 | 13
Anorexia (Metabolism and nutrition disorders) | 2 | 21
Blood albumin decreased (Metabolism and nutrition disorders) | 2 | 20
Hyperglycemia NOS (Metabolism and nutrition disorders) | 3 | 18
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 14
Hyponatremia (Metabolism and nutrition disorders) | 2 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 20
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 27
Taste disturbance (Nervous system disorders) | 0 | 12
Depression NEC (Psychiatric disorders) | 3 | 14
Libido decreased (Psychiatric disorders) | 28 | 23
Dysuria (Renal and urinary disorders) | 42 | 54
Hematuria present (Renal and urinary disorders) | 7 | 16
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 92 | 84
Renal/GU-Other (Renal and urinary disorders) | 8 | 15
Urinary frequency (Renal and urinary disorders) | 118 | 133
Urinary retention (Renal and urinary disorders) | 16 | 14
Gynaecomastia (Reproductive system and breast disorders) | 17 | 38
Impotence (Reproductive system and breast disorders) | 103 | 100
Late RT Toxicity: Other GU: NOS (Reproductive system and breast disorders) | 52 | 45
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 48
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 5 | 12
Menopausal symptoms (Vascular disorders) | 154 | 154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.